CLINICAL TRIAL: NCT01221974
Title: Use of Essure® Micro-inserts in Women With Hydrosalpinx Prior to In Vitro Fertilization: A Prospective, Multicenter, International Feasibility Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Reproductive Science Center (Industry)
Collaborators: Shady Grove Fertility (Unknown)
Responsible Party: Donald Galen M.D., Reproducitve Science Center
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: IVF1
Record Dates: First submitted 2010-10-04; First posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-10

CONDITIONS: Women Who Suffer From Hydrosalpinx That is Causing Infertility and Whom Want a Safer Way of Treamtent
Keywords: Hydrosalpinx or infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Essure,Hydrosalpinx, Infertility (Experimental)
  Interventions: Device: Essure Micro Insert

INTERVENTIONS:
Device: Essure Micro Insert

SUMMARY:
The purpose of this study is to gather safety data related to the use of Essure® micro-inserts in women with hydrosalpinx prior to in vitro fertilization and during pregnancy and to collect data with regard to implantation rates, clinical pregnancy rates, and pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

Women age 21-38 (unless women in ovum donor cycle then age will be included up to 43) who:

Are willing to participate in this clinical study Are able to comprehend and give informed consent for participation in this study Have read, understood and signed an informed consent form Have been unable to achieve pregnancy after trying for 1 year or greater and who have unilateral or bilateral hydrosalpinges as evidenced by laparoscopy or ultrasound or HSG Have a Day #3 serum FSH<10, and Day #3 Estradiol<80 Recipient women undergoing a ovum donor cycle the donor must have a Day 3 serum FSH < 10 and Day 3 Estradiol < 80 Have an antral follicle count 10 or greater for both ovaries combined, if women using ovum donor (follicle count) will be based on eligible donor Have a desire to receive treatment for their HS Are willing to undergo a hysterosalpingogram (HSG) 3 months after Essure placement to confirm proximal tubal occlusion

Exclusion Criteria:

Active or recent upper or lower pelvic infection Known hypersensitivity to nickel as confirmed by skin test Known allergy to contrast media Pregnancy or suspected pregnancy Delivery or termination of pregnancy less than six weeks prior to Essure micro-insert placements BMI > 35 Abnormal pap smear (CIN2 or greater abnormality) within the past year Pelvic malignancy Severely retroverted uterus Evidence of intrauterine abnormalities such as submucous fibroids, polyps, intrauterine adhesions or presence of a uterine septum Abnormal Clomid Challenge Test or abnormal lab values on Day #3 serum FSH and Estradiol Antral follicle count less than 10 (both ovaries combined) Poor general or gynecologic health Inability or refusal to provide informed consent

-

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-07; Primary Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Science Center, San Ramon, California, United States